CLINICAL TRIAL: NCT03685994
Title: The Incidence of Sleep Disorders After Transjugular Intrahepatic Portosystemic Shunt
Brief Title: Sleep Disorders After TIPS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, luo xuefeng, Clinical Professor, West China Hospital
Other Study IDs: SD-TIPS
Record Dates: First submitted 2018-09-23; First posted 2018-09-26 (Actual); Last update posted 2019-04-22 (Actual); Status verified 2019-04

CONDITIONS: Sleep Disorder
MeSH Terms: conditions — Sleep Wake Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- the patients who will undergo TIPS

SUMMARY:
The Purpose of a study to investigate the incidence of postoperative sleep disorders in patients undergoing transjugular intrahepatic portosystemic shunt ,and to analyze the relationship between risk factors and prognosis of sleep disorders.

ELIGIBILITY:
Inclusion Criteria:

1. History of cirrhosis (clinical or by liver biopsy)
2. Portal hypertension patients with defined indications for TIPS treatment
3. Aged 18-75 years old
4. Signed written informed consent

Exclusion Criteria:

1. mental or nervous system diseases
2. Patients with alcoholic cirrhosis who are still drinking
3. Accompanied by serious heart, lung, brain and kidney diseases
4. Preoperative diagnosis of sleep disorder
5. Patients who are illiteracy
6. The total score of the preoperative Hamilton anxiety scale was greater than or equal to 14 points, and the total score of 17 points of the Hamilton depression scale was greater than or equal to 18 points

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 100 patients who underwent TIPS in our hospital due to cirrhosis and portal hypertension.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-08-31 (Actual); Primary Completion 2019-08 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
The incidence of sleep disorders after TIPS | 1 year
  The number of patients who suffer from sleep disorders after TIPS

SECONDARY OUTCOMES:
Incidence of hepatic encephalopathy | 1 year
  The number of patients who suffer from hepatic encephalopathy
mortality | 1 year
  The number of patients who died

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital, Chengdu, Sichuan, China

REFERENCES:
- [Derived] Zhao M, Yan Y, Wang X, Liu B, Luo X. Sleep disturbance in patients with cirrhosis and transjugular intrahepatic portosystemic shunt. BMC Gastroenterol. 2024 Oct 28;24(1):381. doi: 10.1186/s12876-024-03470-x. PMID 39465397